CLINICAL TRIAL: NCT02985060
Title: Mild Hypothermia After Endovascular Treatment in Acute Ischemic Stroke; Prospective, Open, Randomized, Multicenter Phase II Study
Brief Title: Mild Hypothermia After Endovascular Treatment in Acute Ischemic Stroke
Acronym: HELMET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bard Medical Division C.R. Bard Inc (Unknown)
Responsible Party: Principal Investigator, Moon Ku Han, proffessor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELMET ver1.1
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Ischemic Stroke; Thrombolytic Therapy
Keywords: Therapeutic hypothermia
MeSH Terms: conditions — Ischemic Stroke | interventions — Hypothermia, Induced; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic hypothermia group (Experimental): Therapeutic hypothermia using surface cooling device (Arctic Sun) Stroke care based on international guidelines except therapeutic hypothermia using surface cooling device (Arctic Sun)
  Interventions: Device: Arctic Sun; Drug: Saline
- Control group (Other): Stroke care based on international guidelines
  Interventions: Other: Standard treatment

INTERVENTIONS:
Device: Arctic Sun — 1. Induction phase: At a temperature of 4℃, a saline 500 mL or 1 L is intravenously administered.
     Arctic sun (surface freezing equipment) Target temperature: 35±0.5℃ Within 12 hours of the onset of symptoms, the therapeutic hypothermia is performed
  2. Maintenance phase:The use of bedside shivering assessment scale (BSAS) The use of Columbia anti-shivering protocol,Maintenance period: 48 hours
  3. Recovery phase:Rewarming velocity: 0.05~0.1℃ (within 30 hours)
  Other Names: Therapeutic hypothermia
  Arms: Therapeutic hypothermia group
Other: Standard treatment — 1. All the patients receive standard treatment modalities for stroke, which are applicable to the international treatment guidelines.
  2. In all the patients, neurological assessments and NIHSS scoring are performed on a daily basis for 4 days with the help of board-certified nurses or specialists in stroke.
  3. Blood pressure, respiratory rate and heart rate are measured at least once at a 4-hour interval for 4 days.
  4. Using an esophageal thermometer, the central temperature is measured at a 2-hour interval for 5 days.
  Arms: Control group
Drug: Saline
  Arms: Therapeutic hypothermia group

SUMMARY:
To study safety and feasibility of mild therapeutic hypothermia after successful recanalization by mechanical endovascular treatment in patients with acute ischemic stroke and proximal arterial occlusion.

DETAILED DESCRIPTION:
The current clinical trial is an investigator-initiated one, and it is conducted under the multi-center, randomized, open-label, prospective design. The subjects meeting inclusion/exclusion criteria will be assigned to the treatment group or the control group. The randomization ratio is 1:1. The subjects of the treatment group will receive a 2-day hypothermia therapy followed by the process of recovery of temperature within 30 hours (the recovery phase). After 3 months of the onset of symptoms, mRS scores are measured. This is followed by the closure of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who submitted a written informed consent prior to the participation in the current clinical trial (If the subjects have conditions that they cannot decide on study participation according to their own will, they would participate in the study after their legal representatives submitted a written informed consent form. During the period of study participation, if patients' medical conditions are improved, the written informed consent should be submitted again.)
2. Patients with ischemic stroke attributed to carotid artery or middle cerebral artery occlusion achieved successful recanalization (TICI 2b or 3) immediately after endovascular treatment within 8 hours of symptom onset: Onset time was defined as the time when patients were lastly seen normal.
3. Patients of both sexes aged between 18 and 80 years old
4. NIHSS scores of 6-25 points at screening
5. mRS 1 prior to the onset of disease, with proximal cerebral artery occlusion (e.g., those with middle cerebral or internal carotid artery)

Exclusion Criteria:

1. No evaluation for cranial artery before endovascular treatment
2. Patient with emergent stenting insertion in intracranial or extracranial artery
3. Transient ischemic attack or lacunar infarction
4. Platelet counts < 75,000/mm3
5. coagulopathy (INR spontaneously >1.5)
6. Hemodynamic instability
7. acute myocardial infarction, acute unstable angina or severe cardiac failure (NYHA classification ≥III)
8. Sepsis
9. Pregnant or breastfeeding women
10. Premorbid modified Rankin Scale Scores of > 2 points
11. Hypersensitivity or allergy to following: buspirone, dexmedetomidine, meperidine
12. Intracranial hemorrhage or hemorrhagic transformation in initial CT scan
13. Brain tumor or CNS infection
14. Patients who participated in other clinical trials within 3 months
15. Life expectancy within 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome | 3 months after symptom onset
  modified Rankin Scale of 0-2 points at 3 months
mortality at 3 months | 3 months after symptom onset
  mortality at 3 months

SECONDARY OUTCOMES:
Improvements in neurological functions | Volume change on diffusion lesion at 5~7 days
  Changes in the cerebral infarction lesions at 5~7 days
Symptomatic cerebral hemorrhage | within 5~7 days of symptom onset
  deterioration in the National Institute of Health Stroke Scale score of ≥4 points with parenchymal hematoma type 2 documented by CT or MR image

CONTACTS AND LOCATIONS:
Overall Officials: MOON-KU HAN, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang, Seongnam, Gyeoinggido, South Korea

REFERENCES:
- [Derived] Jeong JH, Hong JH, Sohn SI, Park H, Chang JY, Yum KS, Kang J, Han MK. Mild Hypothermia After Endovascular Treatment for Acute Ischemic Stroke: A Pilot Randomized Controlled Trial. Stroke. 2025 Nov;56(11):3100-3107. doi: 10.1161/STROKEAHA.124.049762. Epub 2025 Aug 12. PMID 40791183